CLINICAL TRIAL: NCT00025194
Title: A Phase I And Randomized Phase 2 Trial Of Epothilone B Analogue BMS 247550 (NSC # 710428) Administered Every 21 Days With Or Without Oral Estramustine Phosphate In Patients With Androgen Independent Prostate Cancer
Brief Title: Ixabepilone With or Without Estramustine in Treating Patients With Progressive Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068935; MSKCC-01064; MSKCC-01064A; NCI-3634
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; ixabepilone

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ixabepilone and estramustine, use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether BMS-247550 is more effective with or without estramustine in treating prostate cancer.

PURPOSE: This randomized phase I/II trial is studying the best dose of ixabepilone when given together with estramustine and to see how well giving ixabepilone together with estramustine works compared to ixabepilone alone in treating patients with progressive prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of ixabepilone combined with estramustine in patients with progressive androgen-independent adenocarcinoma of the prostate. (Phase I)
* Compare the safety and efficacy of ixabepilone with or without estramustine in this patient population. (Phase II)
* Correlate the clinical outcomes with reverse transcriptase-polymerase chain reaction-based assay for prostate-specific antigen mRNA in patients treated with these regimens.

OUTLINE: This is a dose-escalation study of ixabepilone (phase I) followed by a randomized, multicenter study (phase II).

* Phase I: Patients receive ixabepilone IV over 3 hours on day 2 and oral estramustine 3 times daily on days 1-5. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of ixabepilone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive ixabepilone IV over 3 hours at the MTD on day 2 and estramustine as in phase I.
  * Arm II: Patients receive ixabepilone IV over 3 hours at the MTD on day 1. Treatment in both arms repeats as in phase I.

Patients are followed every 12 weeks until disease progression.

PROJECTED ACCRUAL: A total of 3-12 patients will be accrued for phase I of this study and a total of 44-92 patients (22-46 per treatment arm) will be accrued for phase II of this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Must have disease progression meeting 1 of the following criteria:

  * Rising prostate-specific antigen (PSA) on at least 3 consecutive measurements taken more than 1 week apart
  * Measurable disease, defined as new or progressive soft tissue masses on CT scan or MRI
  * New metastatic lesions by radionuclide bone scan
* The most recent PSA must be at least 4 ng/mL if no measurable disease is present
* Ineligible if sole manifestation of progressive disease is an increase in disease-related symptoms
* Serum testosterone no greater than 50 ng/mL
* One of the following therapies for maintenance of castrate status required:

  * Must continue on gonadotropin-releasing hormone analogs (e.g., leuprolide or goserelin) to maintain castrate levels of serum testosterone

    * Developed disease progression after discontinuation of the antiandrogen that was part of the first-line hormonal therapy
  * Prior surgical orchiectomy
* Developed disease progression after discontinuation of megestrol
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No history of bleeding disorder that would preclude anticoagulation with warfarin

Hepatic:

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal (ULN)
* PT/PTT normal (unless anticoagulated for other reasons [e.g., atrial fibrillation])

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No significant cardiovascular disease
* No symptomatic congestive heart failure
* No New York Heart Association class III or IV heart disease
* No active unstable angina pectoris
* No cardiac arrhythmia
* No myocardial infarction within the past 6 months
* No history of hemorrhagic or thrombotic cerebrovascular accident or deep venous thrombosis within the past 6 months

Pulmonary:

* No pulmonary embolism within the past 6 months

Other:

* Fertile patients must use effective contraception
* No history of allergic reactions to compounds of similar chemical or biological composition to the epothilones
* No history of recent gastrointestinal bleeding that would preclude anticoagulation with warfarin
* No other concurrent active malignancy except nonmelanomatous skin cancer

  * Disease not considered currently active if completely treated with less than a 30% risk for relapse
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent routine filgrastim (G-CSF) or sargramostim (GM-CSF) except for neutropenic fever
* No concurrent immunotherapy

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* No prior palliative radiotherapy to more than 25% of bone marrow
* No prior radioisotope therapy with strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium
* No concurrent therapeutic radiotherapy
* Concurrent focal radiotherapy for palliation of bone disease-related symptoms allowed at the investigator's discretion

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior major surgery

Other:

* No other concurrent anticancer investigational or commercial agents or therapies
* No concurrent herbal, alternative, or food supplements (e.g., PC-SPES, saw palmetto, or St. John's Wort)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No initiation of bisphosphonates immediately before or during study
* Concurrent bisphosphonates allowed if developed disease progression while on stable doses
* Concurrent daily multivitamin allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Galsky MD, Small EJ, Oh WK, Chen I, Smith DC, Colevas AD, Martone L, Curley T, Delacruz A, Scher HI, Kelly WK. Multi-institutional randomized phase II trial of the epothilone B analog ixabepilone (BMS-247550) with or without estramustine phosphate in patients with progressive castrate metastatic prostate cancer. J Clin Oncol. 2005 Mar 1;23(7):1439-46. doi: 10.1200/JCO.2005.09.042. PMID 15735119
- [Result] Smaletz O, Galsky M, Scher HI, DeLaCruz A, Slovin SF, Morris MJ, Solit DB, Davar U, Schwartz L, Kelly WK. Pilot study of epothilone B analog (BMS-247550) and estramustine phosphate in patients with progressive metastatic prostate cancer following castration. Ann Oncol. 2003 Oct;14(10):1518-24. doi: 10.1093/annonc/mdg415. PMID 14504052
- [Result] Smaletz O, Kelly WK, Horse-Grant D, et al.: Epothilone B analogue (BMS-247550) with estramustine phosphate (EMP) in patients (pts) with progressive castrate-metastatic prostate cancer (PC). [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-732, 184a, 2002.